CLINICAL TRIAL: NCT06734598
Title: Efficacy of Botox Injection of the Masticatory Muscles in Head &Neck Cancer Patients with Trismus After Radiotherapy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202410133MINA
Record Dates: First submitted 2024-12-09; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Trismus; Head and Neck Cancer; Radiation Therapy Recipient; BOTOX
MeSH Terms: conditions — Trismus; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botox injection (Experimental)
  Interventions: Drug: Echo-guided Botox injection
- Normal Saline Injection (Placebo Comparator)
  Interventions: Procedure: echo-guided normal saline injection

INTERVENTIONS:
Drug: Echo-guided Botox injection — Echo-guided Botox injection to the masticatory muscles
  Arms: Botox injection
Procedure: echo-guided normal saline injection — echo-guided normal saline injection
  Arms: Normal Saline Injection

SUMMARY:
Trismus is a common side effect in head and neck cancer patients after radiation therapy. This project aims to explore the therapeutic effect of Botulinum toxin (Botox) injection to the masticatory muscles in the above-mentioned patients.

In this project, Botulinum toxin will be injected into the masticatory muscles (medial pterygoid and masticatory muscles), combined with oral rehabilitation exercises, to reduce the patient's masticatory muscle tension and spasm. Patient's mouth opening range, quality of life, trismus condition and pain will be evaluated to understand its efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18 years old;
2. Head and neck cancer patients must have completed radiotherapy for at least 3 months;
3. Those whose mouth-opening distance is less than or equal to 3.5 cm (the functional cut-off point of trismus) and who have tightness or pain in the masticatory muscles;
4. Medical condition is stable;

Exclusion Criteria:

1. Those who have undergone surgery on their masticatory muscles;
2. Patients with obvious muscle atrophy or complete fibrosis of masticatory muscles ;
3. Those with tumor recurrence at the time of admission;
4. Those whose vital signs are unstable due to acute illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Maximal Incisal Opening | From enrollment to the end of treatment at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No